CLINICAL TRIAL: NCT03525769
Title: Screening With FibroTouch for Advanced Liver Fibrosis in NAFLD Patients With Underlying Type 2 Diabetes：A Registry and Diagnostic Cohort Study
Brief Title: Screening With FibroTouch for Advanced Liver Fibrosis in NAFLD Patients With Underlying Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 007
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes Mellitus; Nonalcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5mL peripheral blood placed in sodium citrate vacuum tube, 5mL peripheral blood serum, and 10mL random urine are collected at the baseline information and specimen collection. 10mL random urine is collected at each time follow-up. All these samples are used for screening potential indicators to evaluate prognosis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetes Mellitus
  Interventions: Diagnostic Test: FibroTouch

INTERVENTIONS:
Diagnostic Test: FibroTouch — FibroTouch is a non-invasive image-guided integrated detection system, providing an integrated detection and comprehensive evaluation program for hepatic fibrosis and hepatic steatosis.
  The FibroTouch is a completely non-invasive liver testing device that can obtain the following results: 1. Liver Fibrosis: quantitative results of hepatic fibrosis; 2. Fatness: quantitative result of hepatic steatosis; 3. Liver tissue morphology: detected by ultrasound imaging.

SUMMARY:
This study is aimed at calculating the incidence of nonalcoholic fatty liver disease (NAFLD), non- alcoholic steatohepatitis (NASH) cirrhosis and advanced fibrosis in patients with type 2 diabetes in China, evaluating the diagnostic efficacy of FibroTouch for hepatic steatosis and fibrosis in these patients, analyzing the long-term prognosis and screening potential risk factors in patients with both type 2 diabetes and NAFLD.

This study will use FibroTouch to screen NAFLD, NASH cirrhosis and advanced fibrosis in patients with type 2 diabetes, compare the results with liver tissue biopsy to assess the clinical value of FibroTouch for the screening of NAFLD in diabetics, then investigate the clinical significance of FibroTouch in assessing the long-term prognosis of patients with diabetes and NAFLD in a prospective cohort, screen risk factors for diabetes with NAFLD and advanced fibrosis.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, observational cohort study. We plan to include 10,000 patients with type 2 diabetes, and use FibroTouch to screen for NAFLD, NASH cirrhosis and advanced fibrosis in these patients. In the group of patients who experienced liver biopsies in clinical practice, we compare their FibroTouch results and liver biopsy pathology results, to evaluate the clinical value of FibroTouch in diagnosing NAFLD, NASH cirrhosis and advanced fibrosis in diabetics. We will calculate the incidence and analyze risk factors of NAFLD, NASH cirrhosis and advanced fibrosis in patients with type 2 diabetes. All patients will be followed-up for 5 years (once a year for patients without cirrhosis, twice a year for patients with cirrhosis), to observed endpoint events. This study will explore the significance of FibroTouch result and other clinical indicators in assessing the long-term prognosis of diabetic patients with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed as type 2 diabetes mellitus(fulfill at least one of the followings):

1. Random plasma glucose levels ≥11.1 mmol/L (twice or more on different days, or once with typical symptoms of diabetes);
2. Fasting plasma glucose levels ≥ 7.0 mmol/L (twice or more on different days, or once with typical symptoms of diabetes);
3. 2h plasma glucose level ≥11.1 mmol/L(twice or more on different days, or once with typical symptoms of diabetes);
4. Previously diagnosed as type 2 diabetes mellitus, plasma glucose level is normal under the current diabetes treatment.

Exclusion Criteria:

* Type 1 diabetes or other types of diabetes;
* Acute or chronic infection;
* Other diseases that cause secondary diabetes: such as pancreatic disease, Cushing's syndrome, acromegaly, glucagonoma, pheochromocytoma, hyperthyroidism, somatostatin, aldosteronoma, etc.;
* Using drugs that cause secondary diabetes (glucocorticoid, thyroid hormone, phenytoin, alpha-interferon, etc.)
* Hepatitis B surface antigen positive (HBsAg+), or hepatitis C antibody positive (Anti-HCV+), or other liver diseases such as alcoholic liver disease;
* Alcohol intake ≥140g/week for men (or ≥70 g/week for women);
* Diagnosed with HCC or other malignancy (in accordance with the appropriate diagnostic criteria);
* Drugs secondary to fatty liver (tamoxifen, amiodarone, valproate, methotrexate, glucocorticoids, etc.).
* During pregnancy or breastfeeding;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study include 10000 type 2 diabetes patients (both inpatients and outpatients of these cooperative member hospitals). We exclude the patients with other type of diabetes, other liver diseases, pregnancy or breastfeeding,malignancy, using the drugs that would possibly cause secondary diabetes or fatty liver.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-05-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | 5 years
  Noticed death of patient at follow-up visit

SECONDARY OUTCOMES:
Liver steatosis | 5 years
  Liver steatosis detected by FibroTouch, or liver biopsy
Advanced fibrosis, compensated cirrhosis, decompensated cirrhosis | 5 years
  Advanced fibrosis, compensated cirrhosis, decompensated cirrhosis detected by FibroTouch, ultrasound, CT, MRI or liver biopsy
Hepatocellular carcinom | 5 years
  Hepatocellular carcinoma detected by CT, MRI or liver biopsy

OTHER OUTCOMES:
Cardiovascular and cerebrovascular diseases | 5 years
  Diagnosed by cardiologists or neurologist
Extrahepatic tumors | 5 years
  Diagnosed by oncologists
Chronic kidney disease | 5 years
  Diagnosed by nephrologists

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Han W, Huang C, Ji Y, Zhou L, Chen J, Hou J. Alterations in the Gut Microbiota and Hepatitis-B-Virus Infection in Southern Chinese Patients With Coexisting Non-Alcoholic Fatty Liver Disease and Type-2 Diabetes Mellitus. Front Med (Lausanne). 2021 Dec 21;8:805029. doi: 10.3389/fmed.2021.805029. eCollection 2021. PMID 34993216